CLINICAL TRIAL: NCT05423002
Title: Mechanisms of Cone Photoreceptors Contribution on Human Neuroendocrine Physiology and Pupillary Light Responses
Brief Title: Effect of Different Color Lights on the Internal Clock and Alertness in Humans
Acronym: CONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Basel (Other)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Principal Investigator, Fatemeh Fazlali, Investigator, University of Basel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ID 2022-00401
Record Dates: First submitted 2022-06-07; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Light Flashing
Keywords: Flickering light; Photoreceptors; Cones
MeSH Terms: conditions — photopsia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Dim light condition as a baseline
  Interventions: Other: Dim light
- Modulation (Active Comparator): Flickering light will be added sinusoidally onto the background light.
  Interventions: Other: Flickering light stimuli
- Background (Sham Comparator): Constant light with maximum half irradiance (50%) of all primaries.
  Interventions: Other: Constant light stimuli

INTERVENTIONS:
Other: Flickering light stimuli — The intervention will be exposed to flickering lights (≤200 lux). More specifically, the participants will be asked to be exposed to a specified flickering light (1Hz, 30 seconds On, and 30 seconds OFF) for 2 hours starting at their habitual bedtime (HBT).
  Arms: Modulation
Other: Constant light stimuli — The intervention will be exposed to constant background lights (≤200 lux). The participants will be asked to be exposed to a specified constant light for 2 hours starting at their habitual bedtime (HBT).
  Arms: Background
Other: Dim light — This light condition is the baseline (≤10 lux).
  Arms: Control

SUMMARY:
The main aim of this study is to investigate the effects of cone-modulated light emitted from a visual display on human circadian physiology and cognitive performance in the evening.

DETAILED DESCRIPTION:
The investigators will generate single/multiple cone-isolating contrasts with equivalent stimuli for other cones and melanopsin photoreceptors. The investigators will assess melatonin suppression under three different light scenarios generated using the method of silent substitution by tuning the spectral composition of the light primaries (e.g. LEDs) such that a single target photoreceptor class is maximally stimulated compared to an equal stimulation of the remaining photoreceptors. Additionally, The investigators will examine pupil response, subjective sleepiness, psychomotor vigilance, visual comfort, and skin temperature under three different light scenarios. This allows for new insights into the lights' cone-contribution mechanism to neuroendocrine physiology in the human retina.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 35 years
* Sex: male or female normal color vision, male dichromat (i.e. tested by CCT, HRR, Farnsworth Munsell 100 Hue Test)
* BMI: 18.5 - 29.9 self-reported weight and height (i.e. normal and overweight according to WHO)
* Signed consent form of participants
* Chronotype: Morningness-Eveningness Questionnaire (31 - 69)
* Sleep Quality: Pittsburgh Sleep Quality Index, PSQI (≤5)

Exclusion Criteria:

* High myopia (> -6 diopters)
* High hyperopia (< +6 diopters)
* Transmeridian travel (>2 time zones) <1 month prior to the first session of the study
* Shift work <3 months prior to the beginning of the study
* Ophthalmological or optometric conditions (cataract, glaucoma, retinal detachment, macular conditions, chronic inflammations, eye injuries, or operations)
* General health concerns or disorders, including heart and cardiovascular, neurological, nephrological, endocrinological, and psychiatric conditions
* Medication impacting on visual, neuroendocrine, sleep, and circadian physiology
* For females only: pregnancy, use of hormonal contraceptives, lactation or breastfeeding
* Drug (urinary drug screening) and alcohol use
* Non-compliance with sleep-wake times: >1 deviation from ±30 minute window sleep and wake-up time
* Extreme chronotype (Munich Chronotype Questionnaire <2 or >7)
* Current participation in other clinical trials

Exclusion criteria due to study requirements:

* Inability to understand and/or follow study materials or procedures
* Insufficient knowledge of project language

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Melatonin concentration | 1 year
  The saliva samples will be collected from participants every 30 min. The investigators hypothesize that the cone flickering light stimuli will have a different melatonin-attenuating effect than the constant background stimuli and that both will have a different effect than baseline.

SECONDARY OUTCOMES:
Vigilance performance | 1 year
  Sustained attention performance will be assessed throughout the study, using an auditory psychomotor vigilance test (PVT) approach. The investigators hypothesize that the flickering light stimuli will produce different reaction times as measured with the PVT than constant light and baseline. Besides, the baseline will not yield the same reaction times as constant background light.
Subjective sleepiness | 1 year
  The investigators will collect subjective sleepiness ratings using the one-question 9-point Karolinska Sleepiness Scale. The investigators hypothesize that sleepiness (ratings) will be different in the flickering light stimuli than in the constant background light and both will be different than baseline.
Visual comfort | 1 year
  To assess each participant's subjective perception of visual comfort, The investigators will use a custom 7-point rating scale that probes brightness, light color, and glare perception based on a selection of questions. The investigators hypothesize that visual discomfort ratings will change in the flickering light stimuli in comparison to the constant background stimuli and baseline.
Skin temperature | 1 year
  The investigators will monitor skin temperatures using six surface temperature thermocouples (BS 1922L Thermochron iButton®, Maxim, US) placed on proximal and distal regions of the body surface. The investigators hypothesize that the temperature of the body skin will be different in the flickering light stimuli than in the constant stimuli and both will have a different effect in comparison to the baseline.
Pupil response | 1 year
  The investigators will measure changes in the pupil area using a silent substitution Pupillograph. The investigators hypothesize that the pupil constriction will be different after exposure to the light conditions as cones and post-receptoral channels adapt to the light stimuli. Besides, the pupil constriction will change differently under the cone-modulated light when the direction of stimuli is identical to the direction of flickering light condition.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Cajochen, Prof, Principal Investigator — Centre for Chronobiology, UPK, University of Basel
Locations (1):
- Centre for Chronobiology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
As the investigators have a plan to submit the study to a registered report journal. The investigators would prefer to share the data after submission.